CLINICAL TRIAL: NCT01180270
Title: Experimental Pilot Trial Assessing Static Graviceptive Function in Patients With Cervical Dystonia
Brief Title: Static Graviceptive Functions in Patients With Cervical Dystonia (CD)
Status: Completed | Type: Observational
Sponsor: Kirsten Elwischger (Other)
Responsible Party: Sponsor-Investigator, Kirsten Elwischger, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: SVV_CD1
Record Dates: First submitted 2010-07-14; First posted 2010-08-12 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Cervical Dystonia
Keywords: Cervical dystonia; torticollis spasmodicus; botulinum toxin; Subjective visual vertical (SVV); SVV; static graviceptive function
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical dystonia: patients suffering from cervical dystonia
  under routine botulinum toxin treatment
- healthy volunteers: control group

SUMMARY:
The purpose of this experimental pilot study is to test the effect of normalization of the head position on the sense of balance at patients with cervical dystonia under routine botulinum toxin treatment.

DETAILED DESCRIPTION:
Background:

The pathophysiological mechanism of cervical dystonia remains unclear. Affection of static graviceptive function has been shown in these patients by measuring the Subjective Visual Vertical (SVV). Healthy subjects, tested with voluntary head tilt, would tilt SVV in the opposite direction of the head. (Müller "E" effect), whereas patients with cervical dystonia set SVV close to true upright with a minimal deviation toward head-tilt. The mechanism of this change in otolith activity in patients with cervical dystonia is still unknown. When treated with botulinum toxin, head deviation will be reversed during a period of approximate 6-9 weeks, with a first peak of action after approximate 3 weeks.

Aim

The aim of this study is to investigate the effect of normalization of the head position under routine intramuscular botulinum toxin application in the cervical muscles (screening, 3 weeks and 9 weeks after injection) on static graviceptive function in patients with cervical dystonia.

Rationale

To our knowledge, the effect of botulinum toxin therapy on static otolith function in patients with cervical dystonia has never been evaluated. This study may provide new informations on the neural plasticity of the vestibular system and may contribute to the understanding of pathophysiological mechanisms of cervical dystonia. Accordingly, it may help developing new treatment strategies for this disease.

Primary hypothesis

There is a difference of at least 6 degrees in subjective visual vertical of patients with CD tested in habitual head position at study inclusion and 3 weeks after injection of Botulinum Toxin.

Study design

Subjective visual vertical will be tested in Patients with CD, who are pre-treated with botulinum toxin and show a good treatment response.

Patients SVV will be assessed before routine botulinum toxin injection (on day of injection), 3 and 9 weeks after injection. For control, SVV will be assessed in normal subjects.

SVV assessment

SVV will be performed by the patient and control while sitting upright in a dark room in different head positions, the head is fixed using a head holder.

In CD patients, SVV will be assessed in different head positions:

1. the habitual head deviation (head deviation will be classified by Tsui score),
2. head fixed in neutral head position (defined as 0° or no head rotation).
3. ear deviated 15° and 30° to ipsilateral and contralateral side, respectively, starting at habitual head deviation

SVV in normal subject, with

A) head fixed in neutral position (defined as 0° or no head rotation),

B) ear deviated 30° to the left,

C) ear deviated 30° to the right,

D) ear deviated 15° to the left,

E) ear deviated 15° to the right, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic CD and willing to participate on the study,
* Isolated laterocollis or laterocollis and torticollis with maximum of 15°rotation
* Aged 18-80 years,
* Under routine treatment with botulinum toxin

Exclusion Criteria:

Patients and Control

* History of vestibular disorders

Patients

* Torticollis with >15°rotation
* Secondary CD (structural MRI lesions, Mb. Wilson)
* Contraindication for intramuscular botulinum toxin therapy: bleeding disorder or anticoagulation therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient botulinum toxin clinic of the department of neurology, medical university of Vienna healthy subjects, residents of vienna
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Subjective visual vertical (SVV), measured in degree (°) | screening
  Assessment: sitting upright in dark room, head is fixed using a head holder with a strap and a neck rest covering the occiput and posterior neck. For deviation of head (0°, 15° and 30° to the left and right side), head holder can be rotated about its midpoint. In front of patient (distance of 100 cm) is dim light bar, which can be rotated about its midpoint by means of an electronic motor and a remote control device. Patients adjust bar for parallel alignment with the perceived gravitational vertical. The operator tilts the bar in a random order 18° from the physical vertical.
SVV in degree (°) | 3 weeks after screeening
  Assessment: sitting upright in dark room, head is fixed using a head holder with a strap and a neck rest covering the occiput and posterior neck. For deviation of head (0°, 15° and 30° to the left and right side), head holder can be rotated about its midpoint. In front of patient (distance of 100 cm) is dim light bar, which can be rotated about its midpoint by means of an electronic motor and a remote control device. Patients adjust bar for parallel alignment with the perceived gravitational vertical. The operator tilts the bar in a random order 18° from the physical vertical.
SVV in degree (°) | 9 weeks after screening
  Assessment: sitting upright in dark room, head is fixed using a head holder with a strap and a neck rest covering the occiput and posterior neck. For deviation of head (0°, 15° and 30° to the left and right side), head holder can be rotated about its midpoint. In front of patient (distance of 100 cm) is dim light bar, which can be rotated about its midpoint by means of an electronic motor and a remote control device. Patients adjust bar for parallel alignment with the perceived gravitational vertical. The operator tilts the bar in a random order 18° from the physical vertical.

SECONDARY OUTCOMES:
Degree of head deviation (°) | screening
  head deviation of patients group in relaxed posture, measured in degrees (°)
degree of head deviation (°) | 3 weeks after screening
  head deviation of patients group in relaxed posture, measured in degrees (°)
degree of head deviation (°) | 9 weeks after screening
  head deviation of patients group in relaxed posture, measured in degrees (°)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Vacherot F, Vaugoyeau M, Mallau S, Soulayrol S, Assaiante C, Azulay JP. Postural control and sensory integration in cervical dystonia. Clin Neurophysiol. 2007 May;118(5):1019-27. doi: 10.1016/j.clinph.2007.01.013. Epub 2007 Mar 23. PMID 17383228
- [Background] Bove M, Brichetto G, Abbruzzese G, Marchese R, Schieppati M. Neck proprioception and spatial orientation in cervical dystonia. Brain. 2004 Dec;127(Pt 12):2764-78. doi: 10.1093/brain/awh291. Epub 2004 Sep 8. PMID 15355873